CLINICAL TRIAL: NCT00955058
Title: Study of Serum Prostatic Specific Antigen (PSA) After Cyproterone Compound Treatment Compared With Oral Contraceptives Pill in Hirsute Polycystic Ovary Syndrome Patients
Brief Title: Evaluation of Serum Prostatic Specific Antigen (PSA) After Cyproterone Compound Treatment Compared With Oral Contraceptives Pill in Hirsute Polycystic Ovary Syndrome Patients
Acronym: PSA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shahid Beheshti University (Other)
Responsible Party: IRHRC, IRRC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSA
Record Dates: First submitted 2009-08-04; First posted 2009-08-07 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PSA; PCO; PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cyproterone compound (Active Comparator): Before and after treatment
  Interventions: Drug: OCP
- oral contraceptive pill (Experimental): Treatment
  Interventions: Drug: OCP

INTERVENTIONS:
Drug: OCP — Daily For 3 months

SUMMARY:
The purpose of this study is to evaluate the effect of oral contraceptive on the serum free prostatic specific antigen (PSA)in women with polycystic ovary syndrome(PCOD)compared with cyproterone compound.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of oral contraceptive on the serum free prostatic specific antigen (PSA)in women with polycystic ovary syndrome(PCOD)compared with cyproterone compound.

This randomized clinical trial included 60 polycystic ovary syndrome patients with hirsutism who were referred to infertility and reproductive health research center and governmental public educational hospital from Feb2007 till Dec 2007. Polycystic ovary syndrome was defined as the diagnostic criteria of 2003 census Rotterdam. Hirsutism was defined as the presence of excessive hair in body and Ferriman -Gallway scores more than 7. Women who received hormone therapy during the last 3 months, on a diet or herbal treatment were excluded from the study. The other exclusion criterion's consisted of Hyperprolactinemia, thyroid disorders, ovarian tumors and Cushing disease. Hirsutism was determined by the Ferriman-Gallway score and recorded for every patient. Blood samples for serum PSA, and the hormonal profile including free testosterone, dehydroepiandrostenedione sulfate(DHEAS) and 17-hydroxyprogesterone(17-OHP) were taken at baseline and at the end of the treatment at the early follicular phase between 3th to 5th days of menstrual cycle at 8 AM. Patients were divided randomly in two treatment groups according to the computer based table. one group received oral contraceptive pills and the other one received cyproterone acetate combined ethinyl-estradiol(Diane) for 3 months. Hirsutism score was evaluated after treatment again. The blood samples were taken during the early follicular phase after 3 months of treatment to avoid pharmacological effect of treatment and serum PSA, free testosterone, DHEAS,17-OHP were measured again. The university ethics committee approved the study and the informed consent was obtained from patients.

ELIGIBILITY:
Inclusion Criteria:

* PCOS patients

Exclusion Criteria:

* Women who received hormone therapy during the last 3 months,
* On a diet
* Herbal treatment
* Hyperprolactinemia
* Thyroid disorders
* Ovarian tumors
* Cushing disease.

Ages: 22 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-02; Primary Completion 2007-02 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Serum free PSA was measured by ultrasensitive chemiluminnicsence enzyme immunoassay | 3 MONTHS

SECONDARY OUTCOMES:
Serum free testosterone was measured by ELISA and 17OHP and DHEAS were measured by radio-immunoassay and gamma scan test. | 3 MONTHS

CONTACTS AND LOCATIONS:
Locations (1):
- Taheripanah, Tehran, Tehran Province, Iran